CLINICAL TRIAL: NCT04449952
Title: Safety and Clinical Efficacy of Mouth Rinses in Type 1 and Type 2 Diabetics: Effect on Oral Soft Tissue, Plaque and Gingivitis
Brief Title: A Study of Mouth Rinses in Type 1 and Type 2 Diabetic Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CCSORC002281; CCSORC002281 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Gingivits in Diabetics
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AFEO-Containing Mouth Rinse (Experimental): Participants with Diabetes (Type 1 and 2) will be randomized to receive AFEO-containing mouth rinse with a marketed fluoride-containing dentifrice, floss (if flossing is part of their normal oral care routine), a marketed soft bristled toothbrush and a timer (if needed). They will brush for at least one minute using full ribbon of a marketed toothpaste on the provided toothbrush. After brushing, rinse for 30 seconds with 20 milliliter (mL) of the assigned mouth rinse twice daily (morning and evening) for 12 consecutive Weeks.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: Alcohol-Free Essential Oil Containing (AFEO) Mouth Rinse Lead Formula; Device: Concept Curve Winter Series Toothbrush; Device: Listerine Cool Mint Floss
- Listerine Cool Mint Mouth Rinse (Marketed product) (Experimental): Participants with Diabetes (Type 1 and 2) will be randomized to receive Listerine cool mint mouth rinse with a marketed fluoride-containing dentifrice, floss (if flossing is part of their normal oral care routine), a marketed soft bristled toothbrush and a timer (if needed). They will brush for at least one minute using full ribbon of a marketed toothpaste on the provided toothbrush. After brushing, rinse for 30 seconds with 20 mL of the assigned mouth rinse twice daily (morning and evening) for 12 consecutive Weeks.
  Interventions: Other: Listerine Cool Mint; Other: Colgate Cavity Protection Toothpaste; Device: Concept Curve Winter Series Toothbrush; Device: Listerine Cool Mint Floss
- 5 Percent (%) Hydroalcohol Mouth Rinse (Experimental): Participants with Diabetes (Type 1 and 2) will be randomized to receive 5% Hydroalcohol mouth rinse with a marketed fluoride-containing dentifrice, floss (if flossing is part of their normal oral care routine), a marketed soft bristled toothbrush and a timer (if needed). They will brush for at least one minute using full ribbon of a marketed toothpaste on the provided toothbrush. After brushing, rinse for 30 seconds with 20 mL of the assigned mouth rinse twice daily (morning and evening) for 12 consecutive Weeks.
  Interventions: Other: 5% Hydroalcohol Mouth Rinse; Other: Colgate Cavity Protection Toothpaste; Device: Concept Curve Winter Series Toothbrush; Device: Listerine Cool Mint Floss

INTERVENTIONS:
Other: Listerine Cool Mint — Participants use 20 mL of Listerine cool mint mouth rinse for 30 sec after brushing
  Arms: Listerine Cool Mint Mouth Rinse (Marketed product)
Other: 5% Hydroalcohol Mouth Rinse — Participants use 20 mL of 5% Hydroalcohol mouth rinse for 30 sec after brushing.
  Arms: 5 Percent (%) Hydroalcohol Mouth Rinse
Other: Colgate Cavity Protection Toothpaste — Participants used Colgate cavity protection toothpaste for brushing teeth twice daily.
Other: Alcohol-Free Essential Oil Containing (AFEO) Mouth Rinse Lead Formula — Participants use 20 mL of AFEO mouth rinse lead formula for 30 sec after brushing.
  Arms: AFEO-Containing Mouth Rinse
Device: Concept Curve Winter Series Toothbrush — Participants will brush teeth at least one minute with provided bristled toothbrush.
Device: Listerine Cool Mint Floss — Participants will use marketed fluoride-containing dentifrice, floss.

SUMMARY:
The purpose of this study is to evaluate mouth rinse formulations for oral soft tissue tolerance and efficacy in plaque/ gingivitis prevention/reduction in Type 1 and Type 2 diabetics when used twice daily as an adjunct to tooth brushing during a twelve-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Adequate oral hygiene (that is brush teeth daily and exhibit no signs of oral neglect)
* Able to comprehend and follow the requirements and restrictions of the study (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical study) based upon research site personnel's assessment
* Negative pregnancy urine tests (females of child bearing potential only)
* Females of childbearing potential must be using a medically-acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the study
* A minimum of 20 gradable teeth including 4 molars with scorable both facial and lingual surfaces.Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, teeth with veneers, or third molars will not be included in the tooth count
* Diabetes Type 1 or Type 2-self reported
* An HB A1C level less than (<) 7.0 percent (%) for Type 1 Diabetes and an HB A1C level of <8.0% for Type 2 Diabetes
* A mean gingival index greater than or equal to (>=) 1.85 per the Modified Gingival Index at Baseline
* A mean plaque index >= 1.95 per the 6 site Turesky modification of the Quigley-Hein Plaque Index at Baseline

Exclusion Criteria:

* Dental prophylaxis within four weeks prior to baseline visit
* More than 3 sites having pocket depths of 5 millimeter (mm) or any sites that are greater than 5 mm in depth
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* A recent history of hypoglycemia requiring medical intervention within the past 30 days
* Use of antibiotics, anti-inflammatory or anticoagulant therapy, phenytoin sodium or diphenylhydantoin, calcium channel blockers, cyclosporin A, immunostimulants/ immunomodulators during the study or within the one month prior to the Baseline exam. Intermittent use of certain anti-inflammatory medication is acceptable at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Whole-Mouth Mean Modified Gingival Index (MGI) Score After 12 Weeks of Product use | 12 Weeks
  Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole Mouth Mean Turesky Plaque Index (TPI) Score After 12 Weeks of Product use | 12 Weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).

SECONDARY OUTCOMES:
Whole Mouth Mean Turesky Plaque Index (TPI) Score After 1 and 6 Weeks of Product use | 1 Week and 6 Weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).
Whole-Mouth Mean Modified Gingival Index (MGI) Score After 6 Weeks of Product use | 6 Weeks
  Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole-Mouth Mean Expanded Bleeding Index (EBI) Score After 6 and 12 Weeks of Product use | 6 Weeks and 12 Weeks
  Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 millimeter (mm) diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).
Percentage of Bleeding Sites, Based on the Expanded Gingival Bleeding Index Score After 6 and 12 Weeks of Product use | 6 Weeks and 12 Weeks
  Percent bleeding sites will be calculated by taking the total number of sites with bleeding score greater than 0 divided by the total number of sites assessed for each participant. Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 millimeter (mm) diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Leite RS, Marlow NM, Fernandes JK, Hermayer K. Oral health and type 2 diabetes. Am J Med Sci. 2013 Apr;345(4):271-273. doi: 10.1097/MAJ.0b013e31828bdedf. PMID 23531957
- [Background] Qaseem A, Wilt TJ, Kansagara D, Horwitch C, Barry MJ, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Fitterman N, Balzer K, Boyd C, Humphrey LL, Iorio A, Lin J, Maroto M, McLean R, Mustafa R, Tufte J. Hemoglobin A1c Targets for Glycemic Control With Pharmacologic Therapy for Nonpregnant Adults With Type 2 Diabetes Mellitus: A Guidance Statement Update From the American College of Physicians. Ann Intern Med. 2018 Apr 17;168(8):569-576. doi: 10.7326/M17-0939. Epub 2018 Mar 6. PMID 29507945
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC002281&attachmentIdentifier=8eb8187b-9c2f-4e13-bb1f-7fc737874806&fileName=Diabetes___CCSORC002281___Final_CSR___Redacted_Version_PDFa.pdf&versionIdentifier=